CLINICAL TRIAL: NCT06306911
Title: Evaluating Kinetics and Bioavailability of Aronia Melanocarpa Extract in Healthy Young and Older Adults
Brief Title: Bioavailability of Aronia Melanocarpa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: BioActor (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BB-BAM
Record Dates: First submitted 2024-02-01; First posted 2024-03-12 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Bioavailability; Kinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aronia Melanocarpa extract (Experimental): a drink consisting of AME (Aronia Melanocarpa extract) and water.
  Interventions: Dietary Supplement: Aronia Melanocarpa extract

INTERVENTIONS:
Dietary Supplement: Aronia Melanocarpa extract — Aronia Melanocarpa extract (AME) consisting of a mixture of anthocyanins and other polyphenols

SUMMARY:
The main objective of this study is to study the bioavailability and kinetics of acute Aronia Melanocarpa supplementation in healthy young (18-35 years) and older adults (55-75 years) adults. During the test day, participants will ingest a drink consisting of Aronia Melanocarpa extract (AME). The bioavailability and kinetics of AME will be assessed via frequent blood sampling, urine collection, and faecal sampling, in which AME and metabolite profiles will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-35 kg/m2
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study

Exclusion Criteria:

* Smoking or smoking cessation < 12 months
* Severe medical conditions, including asthma, kidney failure, auto-inflammatory diseases, rheumatoid arthritis, diabetes mellitus, cardiovascular disease, gastrointestinal disorders such as Crohn's disease, colitis
* Use of dietary supplements or medication affecting the main outcomes of the study (e.g. affecting gut metabolism, blood pressure medication)
* Use of an investigational product within another biomedical intervention trial within the previous month
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Known pregnancy or lactation
* Known allergy to study product
* Difficult venepuncture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Aronia metabolites in blood | time = 0 hours until t = 48 hours
  Concentrations and quality of Aronia metabolites in blood analysed with LC-MS
Aronia metabolites in urine | time = 0 hours until t = 48 hours
  Concentrations and quality of Aronia metabolites in urine analysed with LC-MS

SECONDARY OUTCOMES:
Aronia metabolites in feces | time = 0 hours
  Concentrations and quality of Aronia metabolites in feces analysed with LC-MS
length - baseline characteristics | time = 0 hours
  length
weight - baseline characteristics | time = 0 hours
  weight
blood pressure (systolic and diastolic) - baseline characteristics | time = 0 hours
  blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Prof, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No